CLINICAL TRIAL: NCT06458140
Title: Acute electRophysiOlogical Changes of Ventricular Myocardium Following cArdioneuroablatioN for Asystolic Reflex Syncope
Brief Title: Cardioneuroablation and Ventricular Proarrhythmia
Acronym: Roman4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Prof. Piotr Kulakowski, Professor, Centre of Postgraduate Medical Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16/2024
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Syncope, Vasovagal
Keywords: cardioneuroablation; reflex syncope; ventricular arrhythmia
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardioneuroablation — Radiofrequency ablation of ganglionated plexi of the heart

SUMMARY:
Cardioneuroablation (CNA) is a promising tool to treat patients with asystolic reflex syncope. CNA acts through complete or near complete abolition of vagal nerve chronotropic and dromotropic effects on the heart, resulting in sinus node acceleration and improved atrio-ventricular conduction, which in turn prevents vagally-mediated reflex asystole. However, lack of parasympathetic protection may potentially be proarrhythmic, especially on the ventricular level. Whether this is a real threat is not known. Therefore, the aim of our study is to assess acute effects of CNA-induced total vagal denervation, measured by extracardiac vagal stimulation, on ECG and electrophysiological parameters as well as vulnerability to ventricular arrhythmias. The study group will consist of 50 consecutive patients undergoing CNA in our institution. Cardioneuroablation will be performed in standard manner. The following parameters will be assessed at baseline and after CNA (directly after CNA, after atropine injected after CNA and after isoproterenol bolus injected at the very end of the procedure): QTc interval, QT dispersion, right ventricular action potential duration, right ventricular effective refractory period and susceptibility to complex ventricular arrhythmias using programmed ventricular stimulation.

DETAILED DESCRIPTION:
Cardiac arrhythmias, both atrial and ventricular, can be modulated by changes in autonomic tone. In ventricular arrhythmias, sympathetic tone is thought to be pro-arrhythmic whereas increased parasympathetic tone exerts protective effects. The main mechanisms responsible for parasympathetic protection involve direct effects on ventricular repolarisation, maintaining electrical stability via preservation of gap junction communication between myocytes, reducing heterogeneity of action potential duration, and decreasing circulating catecholamines and inflammatory markers. It has also been shown that enhanced parasympathetic activity increases ventricular fibrillation (VF) threshold. Also, termination of ventricular tachycardia (VT) by manoeuvres leading to augmentation of parasympathetic tone has been demonstrated. Numerous experimental studies showed that vagal nerve stimulation may decrease susceptibility to ventricular arrhythmias.

Cardioneuroablation (CNA) is a new promising method to treat reflex syncope which is due to vagally-induced functional sinus arrest or atrio-ventricular block (AVB). The goal of the procedure is to ablate post-ganglionic endings of parasympathetic part of autonomic nervous system (ANS), located in ganglionated plexi (GP) in the epicardial fat and in the myocardium. Although both sympathetic and parasympathetic nerves are localised in GPs, the latter ones only barely regenerate. Therefore, CNA-induced damage of the parasympathetic part of GP is greater and more durable than that of the sympathetic part of ANS. Because increased vagal activity is one of the main mechanisms leading to reflex sinus arrest or atrio-ventricular (AV) block, targeting this part of ANS by CNA may prevent recurrences of reflex syncope. Indeed, it has been shown that CNA may be effective in approximately 80-90% of very symptomatic subjects with reflex syncope.

While the reduction of parasympathetic drive to the atrial GPs, responsible for sinus node and AV conduction, seems to be logical and effective way for treating hypervagotonic reflex syncope, CNA-induced changes at the ventricular level may be theoretically harmful. As mentioned above, parasympathetic tone exerts protective effects on ventricular arrhythmias. Recently, the long-term safety of CNA has become an issue raised by some investigators. They expressed concerns that CNA-induced chronic and long-lasting decrease in parasympathetic activity may be dangerous during the future life of usually young people undergoing CNA nowadays. For instance, if they develop coronary artery disease, heart failure or other cardiac diseases which increase propensity of ventricular arrhythmias, lack of parasympathetic protection may lead to the occurrence of complex or even life-threatening ventricular arrhythmias.

Data in literature on possible proarrhythmic effects of CNA are limited and not uniform. From the anatomical and physiological point it has been shown many years ago that destruction of cardiac innervation at the atrial level may also damage ventricular innervation downstream. Although CNA targets GP localised mainly around the left and right atria, responsible for sinus and AV nodes innervation, ventricular GPs may be also affected indirectly by alterations in interaction with atrial GPs or even by direct ablation of some of ventricular GPs. According to Pauza et al. there are several ventricular GPs which are located in the epicardial fat surrounding the aortic root, close to right and left coronary artery ostia, at the area of the proximal posterior descending coronary artery, close the proximal right acute marginal coronary artery, and at the origin of the left obtuse marginal coronary artery. However, the number of ventricular GPs is much lower than that of the atrial ones (20% of atrial GPs) and their density is also lower. Thus, it is very likely that during ablation of some "atrial" GPs like postero-medial left GP (PMLGP) or within the coronary sinus (CS) also ventricular GPs integrity and function may be altered.

Specific data in literature on possible pro-arrhythmic effects of CNA on ventricular myocardium are scarce. A few experimental studies suggested that decreasing the parasympathetic drive to the heart by ablating epicardial GP's increases susceptibility to ventricular arrhythmias both in normal and ischaemic animal hearts. Also one recent study showed that acute ischaemia occurring 6 weeks after CNA was associated with significantly higher incidence of VF than in control untreated swine. As far as human data is concerned, a few cases of possible proarrhythmia - polymorphic VT induction after pulmonary vein isolation with concomitant parasympathetic denervation or after pure CNA, have been described.

Susceptibility to complex ventricular arrhythmias before and after institution of pharmacological treatment or performing a procedure can be assessed invasively by measuring drug- or procedure-induced changes in the ventricular effective refractory period (VERP), ventricular action potential duration (VAPD) and directly by using programmed ventricular stimulation (PVS). However, these data in subjects undergoing CNA are lacking.

Apart from invasive measurements, changes in the duration and dispersion of ventricular repolarisation may be indirectly assessed on surface ECG by measuring the corrected QT (QTc) interval and QT dispersion (QTd). Data on the CNA-induced changes on QT are scarce and conflicting. While Aksu et al showed that CNA caused significant shortening of QT interval duration which may be in some situations, such as long QT syndrome, anti-arrhythmic, others showed that PVI with CNA does not change QT interval or that CNA causes prolongation of QT interval which may in fact have proarrhythmic effects. It has also been shown that QTd increases after PVI which is almost always combined with some GPs ablation or after pure CNA. The preliminary results from one excellent CNA centre showed that QTc was significantly prolonged by 25-30 ms immediately after the procedure, only by 5-10 ms one day after CNA, returned to the baseline values 3 months later, and was slightly shorter than at baseline one year after the procedure.

In summary, it is little known about possible proarrhythmic effects of CNA at the ventricular level. This study was set out to explore these effects.

Aim To assess acute effects of CNA-induced total vagal denervation, measured by extracardiac vagal stimulation (ECVS) on ventricular refractoriness and vulnerability to ventricular arrhythmias, in patients undergoing this procedure due to reflex asystolic syncope.

Hypothesis. Acutely, CNA prolongs ventricular effective refractory period, ventricular action potential duration and QT interval without increasing susceptibility to stimulation-induced sustained ventricular arrhythmias. The effects on QTd are difficult to predict.

Methods Patients. The study group will consist of consecutive patients undergoing CNA in our institution. Patients are offered CNA if they have severe, recurrent symptoms due to reflex syncope with ECG documented asystole >3 seconds, especially if associated with injury, or recurrent presyncope with persistent reflex bradycardia. The patients have to have a history of ineffective prior non-pharmacological treatment and positive baseline atropine test (sinus rate acceleration > 30% and no AV block following 2 mg of intravenous atropine). All patients gave informed written consent to undergo CNA and to participate in the study (Ethics Committee approval #33/2024.) Cardioneuroablation. The procedure is performed under general anaesthesia with muscle relaxation using a 3.5 mm irrigated tip catheter (Navistar ThermoCool SmartTouch) with contact force module and electroanatomical system Carto 3 (Biosense Webster, US). The ablation index is set at 500 except coronary sinus (CS) where the target value is 350. Intracardiac echocardiography (ICE) (Acuson SC2000, Siemens, Germany, AcuNav™ Ultrasound Catheter, Biosense Webster, US) is also used throughout the whole procedure and serves for guiding ablation, including identification of presumed GP areas. The extra cardiac vagal stimulation (ECVS) is performed using two diagnostic catheters positioned in the right and left jugular veins utilizing neurostimulator designed by Dr Pachon (Sao Paulo, Brazil) (pulse amplitude of 1 V/kg body weight up to 70 V, 50 ms width, 50 Hz frequency, delivered over 5 sec). Complete bilateral vagal denervation of both sinus and AV nodes (no sinus arrest, slowing of sinus rate no more than 10% compared with baseline and no AV block with PR interval no longer than at baseline), documented on ECVS, is the end-point of CNA.

Ablation is usually started in the left atrium (LA) at the anterior antrum of the right pulmonary vein where the superior paraseptal GP (SPSGP) is located, followed by ablation of the inferior paraseptal GP (IPSGP) at the floor of LA). Next, these GPs are ablated from the right atrium (RA). If the intraprocedural endpoints of CNA are not achieved by ablation of paraseptal GPs, additional applications in the LA at the sites of superior and postero-lateral LA GPs are performed, followed by applications in CS.

At the end of the procedure, atropine test is performed in order to assess the residual, if present, vagal nerve activity. The value of < 10% of increase in sinus rate following atropine injection (2 mg iv) will be taken as successful vagal denervation.

Surface ECG. The QT interval is measured in lead II and corrected for heart rate (QTc) using the Bazett and Fridericia formulas. The QT dispersion (QTd) - the difference between the shortest and the longest QT interval in 12-lead ECG, is also measured. All measurements are performed at baseline and after CNA using electronic callipers (Bard EPLab system) at a speed of 100 mm/sec. The QTc interval is also measured from 12 lead standard ECG at a speed of 25 mm/sec performed one day before and one day after CNA.

Invasive electrophysiology. VAPD will be measured during the procedure before and after CNA from the right ventricle (RV) using unfiltered unipolar recording with contact force (CF) > 10 g, using the same CF value before and after CNA in a given patient. Baseline measurement will be taken just before first RF application at the time when a patient will already be given a full dose of anaesthetic drugs to ensure that all VAPD recordings will be performed under unchanged sedation and muscle relaxation drug regimen. The measurements will be performed during sinus rhythm and during constant atrial pacing at a cycle length of 400 ms and at a speed of 200 mm/sec.

The VERP at baseline and after CNA will be measured during sinus rhythm and after eight-beat drives at cycle length (CL) of 400 ms delivered from the RV. The same protocol will be simultaneously used to perform PVS in order to assess vulnerability to non-sustained VT or sustained VT (lasting >30 sec or causing haemodynamic compromise), polymorphic VT and or VF.

The VAPD, VERP and PVS will be repeated after atropine injection (2 mg) and finally after isoprenaline bolus of 20 mcg at the end of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* severe, recurrent symptoms due to reflex syncope with ECG documented asystole >3 seconds
* history of ineffective prior non-pharmacological treatment
* positive baseline atropine test (sinus rate acceleration > 30% and no atrio-ventricular block following 2 mg of intravenous atropine)
* informed written consent to participate in the study

Exclusion Criteria:

* Lack of consent to participate in the study
* Contraindications to perform right ventricular stimulation

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Inducibility of ventricular arrhythmias | 2 hours
  Programmed ventricular stimulation is used to assess vulnerability to ventricular arrhythmia at baseline and after cardioneuroablation

SECONDARY OUTCOMES:
Corrected QT interval | 2 hours
  Standard ECG is used to assess corrected QT interval before and after cardioneuroablation
QT interval dispersion | 2 hours
  Standard ECG is used to measure QT interval dispersion before and after cardioneuroablation
Right ventricular action potential duration | 2 hours
  Intracardiac ECG recorded from the ablation electrode is used to measure right ventricular action potential duration before and after cardioneuroablation
Effective refractory period of the right ventricle | 2 hours
  During programmed ventricular pacing using eight-beat drive and one extrastimulus delivered at progressively shortened coupling interval is used to assess effective refractory period of the right ventricle before and after cardioneuroablation

CONTACTS AND LOCATIONS:
Overall Officials: Roman Piotrowski, MD PhD, Study Chair — Medical Centre for Postgraduate Education
Locations (1):
- Department of Cardiology, Postgraduate Medical School, Grochowski Hospital, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
On reasonable request from other researchers or other scientific organizations
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available from January 2025 to January 2027
Access Criteria: direct e-mail contact

REFERENCES:
- [Background] Chakraborty P, Chen PS, Gollob MH, Olshansky B, Po SS. Potential consequences of cardioneuroablation for vasovagal syncope: A call for appropriately designed, sham-controlled clinical trials. Heart Rhythm. 2024 Apr;21(4):464-470. doi: 10.1016/j.hrthm.2023.12.004. Epub 2023 Dec 16. PMID 38104955
- [Result] Zhu C, Hanna P, Rajendran PS, Shivkumar K. Neuromodulation for Ventricular Tachycardia and Atrial Fibrillation: A Clinical Scenario-Based Review. JACC Clin Electrophysiol. 2019 Aug;5(8):881-896. doi: 10.1016/j.jacep.2019.06.009. Epub 2019 Aug 19. PMID 31439288
- [Result] Brack KE, Coote JH, Ng GA. Vagus nerve stimulation protects against ventricular fibrillation independent of muscarinic receptor activation. Cardiovasc Res. 2011 Aug 1;91(3):437-46. doi: 10.1093/cvr/cvr105. Epub 2011 May 16. PMID 21576131
- [Result] Pachon JC, Pachon EI, Pachon JC, Lobo TJ, Pachon MZ, Vargas RN, Jatene AD. "Cardioneuroablation"--new treatment for neurocardiogenic syncope, functional AV block and sinus dysfunction using catheter RF-ablation. Europace. 2005 Jan;7(1):1-13. doi: 10.1016/j.eupc.2004.10.003. PMID 15670960
- [Result] Piotrowski R, Baran J, Sikorska A, Krynski T, Kulakowski P. Cardioneuroablation for Reflex Syncope: Efficacy and Effects on Autonomic Cardiac Regulation-A Prospective Randomized Trial. JACC Clin Electrophysiol. 2023 Jan;9(1):85-95. doi: 10.1016/j.jacep.2022.08.011. Epub 2022 Aug 28. PMID 36114133
- [Result] Kulakowski P, Baran J, Sikorska A, Krynski T, Niedzwiedz M, Soszynska M, Piotrowski R. Cardioneuroablation for reflex asystolic syncope: Mid-term safety, efficacy, and patient's acceptance. Heart Rhythm. 2024 Mar;21(3):282-291. doi: 10.1016/j.hrthm.2023.11.022. Epub 2023 Nov 29. PMID 38036236